CLINICAL TRIAL: NCT01340898
Title: Immunogenicity and Safety Study of GSK Biologicals' Meningococcal Conjugate Vaccine (GSK 134612) When Co-administered With Routine Vaccines in Healthy Infants and Toddlers
Brief Title: Immunogenicity and Safety Study of GSK Biologicals' Meningococcal Conjugate Vaccine When Co-administered With Routine Vaccines in Healthy Infants and Toddlers
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 114858; 2013-002537-37 (EudraCT Number)
Record Dates: First submitted 2011-04-14; First posted 2011-04-25 (Estimated); Results first posted 2019-08-06 (Actual); Last update posted 2019-08-06 (Actual); Status verified 2019-06

CONDITIONS: Meningococcal Infection
Keywords: meningococcal conjugate vaccine; serogroups A,C, W-135 or Y; meningococcal diseases; Immunogenicity; Neisseria meningitidis; co-administration; routine vaccines
MeSH Terms: conditions — Meningococcal Infections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Nimenrix 3+1 Group (Experimental): Subjects, male and female, received 4 doses of Nimenrix™ vaccine (3 doses at 2, 4 and 6 months of age followed by a booster dose at 15-18 months of age) and 4 doses of Synflorix™ and Infanrix-IPV/Hiberix™ vaccines (at 2, 4, 6 and 15-18 months of age). All vaccines were administered intramuscularly (IM) in the anterolateral region of the thigh.
  Interventions: Biological: Meningococcal vaccine GSK 134612; Biological: SynflorixTM; Biological: Infanrix-IPV/HiberixTM
- Nimenrix 1+1 Group (Experimental): Subjects, male and female, received 2 doses of Nimenrix™ vaccine (1 dose at 6 months of age followed by a booster dose at 15-18 months of age) and 4 doses of Synflorix™ and Infanrix-IPV/Hiberix™ vaccines (at 2, 4, 6 and 15-18 months of age). All vaccines were administered intramuscularly (IM) in the anterolateral region of the thigh.
  Interventions: Biological: Meningococcal vaccine GSK 134612; Biological: SynflorixTM; Biological: Infanrix-IPV/HiberixTM
- Nimenrix Control Group (Experimental): Subjects, male and female, received 1 dose of Nimenrix™ at 15-18 months of age and 4 doses of Synflorix™ and Infanrix-IPV/Hiberix™ vaccines (at 2, 4, 6 and 15-18 months of age). All vaccines were administered intramuscularly (IM) in the anterolateral region of the thigh.
  Interventions: Biological: Meningococcal vaccine GSK 134612; Biological: SynflorixTM; Biological: Infanrix-IPV/HiberixTM

INTERVENTIONS:
Biological: Meningococcal vaccine GSK 134612 — Intramuscular injection
Biological: SynflorixTM — Intramuscular injection
Biological: Infanrix-IPV/HiberixTM — Intramuscular injection

SUMMARY:
This study evaluates the immunogenicity and safety of the meningococcal conjugate vaccine GSK 134612 in healthy infants, when co-administered with other infant vaccines, on three different dose schedules.

DETAILED DESCRIPTION:
This protocol has been updated following Protocol Amendment 1 date 26 July 2011 leading to the update of enrollment, a secondary outcome measure, intervention and exclusion criteria sections.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that parent(s)/Legally Acceptable Representative(s) [LAR(s)] can and will comply with the requirements of the protocol.
* A male or female, 6 to 12 weeks (42-90 days) of age at the time of the first vaccination.
* Written informed consent obtained from the parent(s)/LAR(s) of the subject.
* Healthy subjects as established by medical history and clinical examination before entering into the study.
* Born after a gestation period of at least 36 weeks.

Exclusion Criteria:

* Child in care.
* Use of any investigational or non-registered product other than the study vaccine(s) within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Extended administration of immunosuppressants or other immune-modifying drugs since birth.
* Planned administration/administration of a vaccine not foreseen by the study protocol during the period 30 days before and after each study vaccine administration, with the exception of rotavirus vaccine and seasonal or pandemic influenza vaccine.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product.
* Previous vaccination against diphtheria , tetanus, pertussis, polio (with the exception of a birth dose of OPV), Haemophilus influenzae type b, Streptococcus pneumonia.
* History of receipt of meningococcal vaccine.
* Subjects who received a birth dose Hepatitis B vaccines within the 30 days before the administration of the first study vaccine.
* History of or intercurrent diphtheria, tetanus, pertussis, polio, Haemophilus influenzae type b disease, pneumococcal and/or meningococcal disease.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination (no laboratory testing required).
* Family history of congenital or hereditary immunodeficiency.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of th

Ages: 6 Weeks to 12 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 753 (Actual)
Dates: Start 2012-01-27 (Actual); Primary Completion 2014-08-04 (Actual); Study Completion 2015-10-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- GSK Investigational Site, Beirut, Lebanon
- GSK Investigational Site, Durango, Mexico

REFERENCES:
- [Derived] Dbaibo G, Tinoco Favila JC, Traskine M, Jastorff A, Van der Wielen M. Immunogenicity and safety of MenACWY-TT, a meningococcal conjugate vaccine, co-administered with routine childhood vaccine in healthy infants: A phase III, randomized study. Vaccine. 2018 Jun 27;36(28):4102-4111. doi: 10.1016/j.vaccine.2018.05.046. Epub 2018 May 18. PMID 29784470

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of 753 subjects enrolled, 3 subjects were not vaccinated and hence not considered to have started the study.
Groups:
- Nimenrix 3+1 Group: Subjects, male and female, received 4 doses of Nimenrix vaccine (3 doses at 2, 4 and 6 months of age followed by a booster dose at 15-18 months of age) and 4 doses of Synflorix and Infanrix-IPV/Hiberix vaccines (at 2, 4, 6 and 15-18 months of age). All vaccines were administered intramuscularly (IM) in the anterolateral region of the thigh.
- Nimenrix 1+1 Group: Subjects, male and female, received 2 doses of Nimenrix vaccine (1 dose at 6 months of age followed by a booster dose at 15-18 months of age) and 4 doses of Synflorix and Infanrix-IPV/Hiberix vaccines (at 2, 4, 6 and 15-18 months of age). All vaccines were administered intramuscularly (IM) in the anterolateral region of the thigh.
- Nimenrix Control Group: Subjects, male and female, received 1 dose of Nimenrix at 15-18 months of age and 4 doses of Synflorix and Infanrix-IPV/Hiberix vaccines (at 2, 4, 6 and 15-18 months of age). All vaccines were administered intramuscularly (IM) in the anterolateral region of the thigh.
Period: Primary Phase
Arm/Group | Nimenrix 3+1 Group | Nimenrix 1+1 Group | Nimenrix Control Group
Started | 376 | 187 | 187
Completed | 360 | 178 | 181
Not Completed | 16 | 9 | 6
Not completed — Serious Adverse Events | 0 | 0 | 1
Not completed — Withdrawal by Subject | 8 | 7 | 5
Not completed — Migrated/moved from study area | 4 | 1 | 0
Not completed — Lost to Follow-up | 4 | 1 | 0
Period: Booster Phase
Arm/Group | Nimenrix 3+1 Group | Nimenrix 1+1 Group | Nimenrix Control Group
Started | 342 | 166 | 170
Completed | 332 | 164 | 163
Not Completed | 10 | 2 | 7
Not completed — Withdrawal by Subject | 3 | 0 | 4
Not completed — Migrated/moved from study area | 3 | 0 | 0
Not completed — Lost to Follow-up | 4 | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nimenrix 3+1 Group | Nimenrix 1+1 Group | Nimenrix Control Group | Total
Number analyzed (Participants) | 376 | 187 | 187 | 750
Age, Continuous [Mean (Standard Deviation); unit: Weeks] | 8.1 (1.6) | 8.1 (1.7) | 8.2 (1.7) | 8.12 (1.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 182 | 105 | 95 | 382
  Male | 194 | 82 | 92 | 368
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White - Arabic / North African Heritage | 199 | 100 | 99 | 398
  White - Caucasian / European Heritage | 1 | 0 | 1 | 2
  Mixed Origin | 176 | 87 | 87 | 350

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Serum Bactericidal Assay Using Rabbit Complement (rSBA) Against Neisseria Meningitidis Serogroups Antibody Titers Greater Than or Equal to (≥) 1:8, One Month Post Dose 3 for the Nimenrix 3+1 Group
Description: The cut-off value for the rSBA titers was ≥ 1:8. Neisseria meningitidis serogroups A, C, W-135, Y (rSBA-MenA, rSBA-MenC, rSBA-MenW-135 and rSBA-MenY) antibodies were assessed.
Time Frame: At Month 5 (one month post-dose 3)
Population: The analysis was performed on the According-to-Protocol (ATP) cohort for immunogenicity adapted for each timepoint, which included all eligible subjects, who complied with the vaccination schedule and for whom data concerning immunogenicity endpoint measures were available. This endpoint was specified to be analysed for the Nimenrix 3+1 Group only.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix 3+1 Group
Number analyzed (Participants) | 328
Participants
  rSBA-MenA | 328
  rSBA-MenC | 327
  rSBA-MenW-135: number analyzed (Participants) | 327
  rSBA-MenW-135 | 325
  rSBA-MenY | 327
Statistical Analysis 1: Comparison: Nimenrix 3+1 Group; Demonstration of the immunogenicity of the Nimenrix™ conjugate vaccine in terms of bactericidal antibodies to N. meningitidis serogroup A one-month post-dose 3 of Nimenrix™ vaccine at 7 months of age in healthy infants; Test type: Superiority or Other; Percentage of subjects = 100, 95% CI 2-sided [98.9 to 100] — Immunogenicity was considered demonstrated if the lower limit of the two-sided exact 95% confidence interval (CI) for the percentage of subjects with rSBA titre ≥ 1:8 was greater than or equal to the pre-defined clinical limit of 80%
Statistical Analysis 2: Comparison: Nimenrix 3+1 Group; Demonstration of the immunogenicity of the Nimenrix™ conjugate vaccine in terms of bactericidal antibodies to N. meningitidis serogroup C one-month post-dose 3 of Nimenrix™ vaccine at 7 months of age in healthy infants; Test type: Superiority or Other; Percentage of subjects = 99.7, 95% CI 2-sided [98.3 to 100] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Nimenrix 3+1 Group; Demonstration of the immunogenicity of the Nimenrix™ conjugate vaccine in terms of bactericidal antibodies to N. meningitidis serogroup W-135 one-month post-dose 3 of Nimenrix™ vaccine at 7 months of age in healthy infants; Test type: Superiority or Other; Percentage of subjects = 99.4, 95% CI 2-sided [97.8 to 99.9] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Nimenrix 3+1 Group; Demonstration of the immunogenicity of the Nimenrix™ conjugate vaccine in terms of bactericidal antibodies to N. meningitidis serogroup Y one-month post-dose 3 of Nimenrix™ vaccine at 7 months of age in healthy infants; Test type: Superiority or Other; Percentage of subjects = 99.7, 95% CI 2-sided [98.3 to 100] — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Number of Subjects With rSBA-MenA, rSBA-MenC, rSBA-MenW-135 and rSBA-MenY Antibody Titers Greater Than or Equal to (≥) 1:8 Prior to and One Month After the Booster Dose for the Nimenrix 3+1 Group
Description: The cut-off value for the rSBA titers was ≥ 1:8
Time Frame: At Month 13 (prior booster) and at Month 14 (one month after the booster dose)
Population: The analysis was performed on the According-to-Protocol (ATP) cohort for immunogenicity adapted for each timepoint, which included all eligible subjects, who complied with the vaccination schedule and for whom data concerning immunogenicity endpoint measures were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix 3+1 Group
Number analyzed (Participants) | 284
Participants
  rSBA-MenA, M13: number analyzed (Participants) | 276
  rSBA-MenA, M13 | 225
  rSBA-MenA, M14: number analyzed (Participants) | 283
  rSBA-MenA, M14 | 283
  rSBA-MenC, M13: number analyzed (Participants) | 276
  rSBA-MenC, M13 | 190
  rSBA-MenC, M14: number analyzed (Participants) | 283
  rSBA-MenC, M14 | 282
  rSBA-MenW-135, M13: number analyzed (Participants) | 257
  rSBA-MenW-135, M13 | 225
  rSBA-MenW-135, M14 | 284
  rSBA-MenY, M13: number analyzed (Participants) | 275
  rSBA-MenY, M13 | 240
  rSBA-MenY, M14 | 284

3. Secondary Outcome: Number of Subjects With rSBA-MenA, rSBA-MenC, rSBA-MenW-135 and rSBA-MenY Antibody Titers Greater Than or Equal to (≥) 1:128, One Month Post-dose 3, Prior to and One Month After the Booster Dose for the Nimenrix 3+1 Group
Description: The cut-off value for the rSBA titers was ≥ 1:128
Time Frame: At Months 5 (one month post-dose 3), 13 (prior booster-dose) and 14 (one month after the booster dose)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix 3+1 Group
Number analyzed (Participants) | 328
Participants
  rSBA-MenA, M5 | 321
  rSBA-MenA, M13: number analyzed (Participants) | 276
  rSBA-MenA, M13 | 146
  rSBA-MenA, M14: number analyzed (Participants) | 283
  rSBA-MenA, M14 | 282
  rSBA-MenC, M5 | 318
  rSBA-MenC, M13: number analyzed (Participants) | 276
  rSBA-MenC, M13 | 93
  rSBA-MenC, M14: number analyzed (Participants) | 283
  rSBA-MenC, M14 | 282
  rSBA-MenW-135, M5: number analyzed (Participants) | 327
  rSBA-MenW-135, M5 | 313
  rSBA-MenW-135, M13: number analyzed (Participants) | 275
  rSBA-MenW-135, M13 | 122
  rSBA-MenW-135, M14: number analyzed (Participants) | 284
  rSBA-MenW-135, M14 | 284
  rSBA-MenY, M5 | 312
  rSBA-MenY, M13: number analyzed (Participants) | 275
  rSBA-MenY, M13 | 121
  rSBA-MenY, M14: number analyzed (Participants) | 284
  rSBA-MenY, M14 | 283

4. Secondary Outcome: rSBA-MenA, rSBA-MenC, rSBA-MenW-135 and rSBA-MenY Antibody Titers One Month Post Dose 3, Prior to and One Month After the Booster Dose for the Nimenrix 3+1 Group
Description: Antibody titers are presented as geometric mean titers (GMTs).
Time Frame: At Months 5 (one month post-dose 3), 13 (prior booster-dose) and 14 (one month after the booster dose)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Nimenrix 3+1 Group
Number analyzed (Participants) | 328
Titers
  rSBA-MenA, M5 | 577.5 [520.7 to 640.6]
  rSBA-MenA, M13: number analyzed (Participants) | 276
  rSBA-MenA, M13 | 71.1 [56.6 to 89.3]
  rSBA-MenA, M14: number analyzed (Participants) | 283
  rSBA-MenA, M14 | 2366.4 [2134.8 to 2623.1]
  rSBA-MenC, M5 | 803.1 [710.4 to 907.8]
  rSBA-MenC, M13: number analyzed (Participants) | 276
  rSBA-MenC, M13 | 33.9 [27.4 to 41.9]
  rSBA-MenC, M14: number analyzed (Participants) | 283
  rSBA-MenC, M14 | 2761.2 [2461.2 to 3097.9]
  rSBA-MenW-135, M5: number analyzed (Participants) | 327
  rSBA-MenW-135, M5 | 1190.3 [1019.3 to 1390.1]
  rSBA-MenW-135, M13: number analyzed (Participants) | 275
  rSBA-MenW-135, M13 | 52.0 [42.2 to 64.2]
  rSBA-MenW-135, M14: number analyzed (Participants) | 284
  rSBA-MenW-135, M14 | 3696.9 [3242.8 to 4214.7]
  rSBA-MenY, M5 | 647.4 [566.6 to 739.6]
  rSBA-MenY, M13: number analyzed (Participants) | 275
  rSBA-MenY, M13 | 66.3 [54.3 to 81.0]
  rSBA-MenY, M14: number analyzed (Participants) | 284
  rSBA-MenY, M14 | 2778.6 [2472.5 to 3122.5]

5. Secondary Outcome: Number of Subjects With rSBA-MenA, rSBA-MenC, rSBA-MenW-135 and rSBA-MenY Antibody Titers Greater Than or Equal to (≥) the Cut-off Values for the Nimenrix 1+1 and Nimenrix Control Groups
Description: The cut-off values for the rSBA antibody titers were ≥ 1:8 and ≥ 1:128
Time Frame: At Months 5 (one month post-primary dose for Nimenrix 1+1 Group), 13 (prior booster dose for Nimenrix 1+1 and prior primary dose for Nimenrix Control Group) and 14 (post booster dose for Nimenrix 1+1 and post-primary dose for Nimenrix Control Group)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix 1+1 Group | Nimenrix Control Group
Number analyzed (Participants) | 163 | 163
Participants
  rSBA-MenA, M5, ≥ 1:8 | 161 | 6
  rSBA-MenA, M13, ≥ 1:8: number analyzed (Participants) | 131 | 132
  rSBA-MenA, M13, ≥ 1:8 | 107 | 19
  rSBA-MenA, M14, ≥ 1:8: number analyzed (Participants) | 139 | 135
  rSBA-MenA, M14, ≥ 1:8 | 138 | 133
  rSBA-MenC, M5, ≥ 1:8: number analyzed (Participants) | 163 | 162
  rSBA-MenC, M5, ≥ 1:8 | 162 | 6
  rSBA-MenC, M13, ≥ 1:8: number analyzed (Participants) | 131 | 132
  rSBA-MenC, M13, ≥ 1:8 | 86 | 3
  rSBA-MenC, M14, ≥ 1:8: number analyzed (Participants) | 139 | 135
  rSBA-MenC, M14, ≥ 1:8 | 138 | 130
  rSBA-MenW-135, M5, ≥ 1:8 | 153 | 4
  rSBA-MenW-135, M13, ≥ 1:8: number analyzed (Participants) | 131 | 132
  rSBA-MenW-135, M13, ≥ 1:8 | 102 | 7
  rSBA-MenW-135, M14, ≥ 1:8: number analyzed (Participants) | 139 | 135
  rSBA-MenW-135, M14, ≥ 1:8 | 139 | 131
  rSBA-MenY, M5, ≥ 1:8: number analyzed (Participants) | 163 | 162
  rSBA-MenY, M5, ≥ 1:8 | 161 | 16
  rSBA-MenY, M13, ≥ 1:8: number analyzed (Participants) | 131 | 132
  rSBA-MenY, M13, ≥ 1:8 | 116 | 24
  rSBA-MenY, M14, ≥ 1:8: number analyzed (Participants) | 139 | 135
  rSBA-MenY, M14, ≥ 1:8 | 139 | 131
  rSBA-MenA, M5, ≥ 1:128 | 155 | 6
  rSBA-MenA, M13, ≥ 1:128: number analyzed (Participants) | 131 | 132
  rSBA-MenA, M13, ≥ 1:128 | 88 | 16
  rSBA-MenA, M14, ≥ 1:128: number analyzed (Participants) | 139 | 135
  rSBA-MenA, M14, ≥ 1:128 | 138 | 132
  rSBA-MenC, M5, ≥ 1:128: number analyzed (Participants) | 163 | 162
  rSBA-MenC, M5, ≥ 1:128 | 151 | 5
  rSBA-MenC, M13, ≥ 1:128: number analyzed (Participants) | 131 | 132
  rSBA-MenC, M13, ≥ 1:128 | 39 | 1
  rSBA-MenC, M14, ≥ 1:128: number analyzed (Participants) | 139 | 135
  rSBA-MenC, M14, ≥ 1:128 | 137 | 128
  rSBA-MenW-135, M5, ≥ 1:128 | 151 | 4
  rSBA-MenW-135, M13, ≥ 1:128: number analyzed (Participants) | 131 | 132
  rSBA-MenW-135, M13, ≥ 1:128 | 65 | 7
  rSBA-MenW-135, M14, ≥ 1:128: number analyzed (Participants) | 139 | 135
  rSBA-MenW-135, M14, ≥ 1:128 | 138 | 131
  rSBA-MenY, M5, ≥ 1:128: number analyzed (Participants) | 163 | 162
  rSBA-MenY, M5, ≥ 1:128 | 159 | 16
  rSBA-MenY, M13, ≥ 1:128: number analyzed (Participants) | 131 | 132
  rSBA-MenY, M13, ≥ 1:128 | 70 | 23
  rSBA-MenY, M14, ≥ 1:128: number analyzed (Participants) | 139 | 135
  rSBA-MenY, M14, ≥ 1:128 | 137 | 131

6. Secondary Outcome: rSBA-MenA, rSBA-MenC, rSBA-MenW-135 and rSBA-MenY Antibody Titers for Nimenrix 1+1 and Nimenrix Control Groups
Description: Antibody titers are presented as geometric mean titers (GMTs).
Time Frame: At Months 5 (one month post-primary dose for Nimenrix 1+1 Group), 13 (prior booster dose for Nimenrix 1+1 and prior primary dose for Nimenrix Control Group) and 14 (post booster dose Nimenrix 1+1 and post-primary dose for Nimenrix Control Group)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Nimenrix 1+1 Group | Nimenrix Control Group
Number analyzed (Participants) | 163 | 163
Titers
  rSBA-MenA, M5, ≥ 1:8 | 1332.9 [1035.2 to 1716.2] | 4.8 [4.1 to 5.5]
  rSBA-MenA, M13, ≥ 1:8: number analyzed (Participants) | 131 | 132
  rSBA-MenA, M13, ≥ 1:8 | 125.3 [84.4 to 186.1] | 7.2 [5.5 to 9.3]
  rSBA-MenA, M14, ≥ 1:8: number analyzed (Participants) | 139 | 135
  rSBA-MenA, M14, ≥ 1:8 | 2762.3 [2310.3 to 3302.8] | 2918.7 [2264.6 to 3761.7]
  rSBA-MenC, M5, ≥ 1:8: number analyzed (Participants) | 163 | 162
  rSBA-MenC, M5, ≥ 1:8 | 591.6 [482.3 to 725.8] | 4.7 [4.1 to 5.4]
  rSBA-MenC, M13, ≥ 1:8: number analyzed (Participants) | 131 | 132
  rSBA-MenC, M13, ≥ 1:8 | 27.4 [20.6 to 36.6] | 4.2 [3.9 to 4.4]
  rSBA-MenC, M14, ≥ 1:8: number analyzed (Participants) | 139 | 135
  rSBA-MenC, M14, ≥ 1:8 | 2525.2 [2102.1 to 3033.3] | 768.1 [593.0 to 995.0]
  rSBA-MenW-135, M5, ≥ 1:8 | 1255.9 [917.0 to 1720.0] | 4.6 [4.0 to 5.2]
  rSBA-MenW-135, M13, ≥ 1:8: number analyzed (Participants) | 131 | 132
  rSBA-MenW-135, M13, ≥ 1:8 | 63.3 [45.6 to 87.9] | 5.0 [4.2 to 5.8]
  rSBA-MenW-135, M14, ≥ 1:8: number analyzed (Participants) | 139 | 135
  rSBA-MenW-135, M14, ≥ 1:8 | 3144.7 [2636.9 to 3750.4] | 5240.7 [3855.5 to 7123.7]
  rSBA-MenY, M5, ≥ 1:8: number analyzed (Participants) | 163 | 162
  rSBA-MenY, M5, ≥ 1:8 | 1469.9 [1186.5 to 1821.0] | 6.3 [5.0 to 7.8]
  rSBA-MenY, M13, ≥ 1:8: number analyzed (Participants) | 131 | 132
  rSBA-MenY, M13, ≥ 1:8 | 106.4 [76.4 to 148.1] | 9.4 [6.8 to 12.9]
  rSBA-MenY, M14, ≥ 1:8: number analyzed (Participants) | 139 | 135
  rSBA-MenY, M14, ≥ 1:8 | 2748.6 [2301.4 to 3282.6] | 4202.5 [3219.9 to 5485.1]

7. Secondary Outcome: Number of Subjects With Booster Responses for rSBA-MenA, C rSBA-MenC, Y rSBA-MenY and W-135 rSBA-MenW-135 in Nimenrix 3+1 and Nimenrix 1+1 Groups and With Vaccine Response in Nimenrix Control Group
Description: Vaccine/Booster response was defined as: for seronegative subjects (rSBA titers < 1:8 pre-vaccination at Month 13), antibody titer ≥ 1:32 at post vaccination; for seropositive subjects (rSBA titers >= 1:8 pre-vaccination at Month 13), antibody titer at post vaccination ≥ 4-fold the pre vaccination antibody titer.
Time Frame: At Month 14 (one month post-booster dose for Nimenrix 3+1 and Nimenrix 1+1 and post-primary dose for Nimenrix Control Group)
Population: The analysis was performed on the Booster According-to-Protocol (ATP) cohort for immunogenicity, which included all eligible subjects, who complied with the vaccination schedule at Month 13 (booster dose for Nimenrix 3+1 and Nimenrix 1+1 and first dose in Nimenrix Control) and for whom data concerning immunogenicity endpoint measures were available
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix 3+1 Group | Nimenrix 1+1 Group | Nimenrix Control Group
Number analyzed (Participants) | 275 | 131 | 132
Participants
  rSBA-MenA | 248 | 108 | 125
  rSBA-MenC | 270 | 129 | 126
  rSBA-MenW-135 | 272 | 122 | 128
  rSBA-MenY | 267 | 121 | 125

8. Secondary Outcome: Number of Subjects With Serum Bactericidal Assay Using Human Complement Against Neisseria Meningitidis Serogroups A, C, W-135, Y Antibody Titers Greater Than or Equal to (≥) the Cut-off Values (One Month Post-primary for Nimenrix 3+1 and 1+1 Groups)
Description: The cut-off value for the hSBA titers was ≥ 1:4 and ≥ 1:8.
Time Frame: At Month 5 (one month post-primary for Nimenrix 3+1 and Nimenrix 1+1 Groups)
Population: The analysis was performed on the According-to-Protocol (ATP) cohort for immunogenicity adapted for each timepoint, which included all eligible subjects for whom data concerning immunogenicity endpoint measures were available. The analysis was performed in a randomized subset of 50% of subjects from each group.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix 3+1 Group | Nimenrix 1+1 Group | Nimenrix Control Group
Number analyzed (Participants) | 147 | 66 | 59
Participants
  hSBA-MenA, ≥ 1:4: number analyzed (Participants) | 136 | 59 | 51
  hSBA-MenA, ≥ 1:4 | 136 | 58 | 9
  hSBA-MenC, ≥ 1:4 | 147 | 66 | 3
  hSBA-MenW-135, ≥ 1:4: number analyzed (Participants) | 107 | 47 | 42
  hSBA-MenW-135, ≥ 1:4 | 107 | 41 | 0
  hSBA-MenY, ≥ 1:4: number analyzed (Participants) | 127 | 52 | 42
  hSBA-MenY, ≥ 1:4 | 127 | 48 | 1
  hSBA-MenA, ≥ 1:8: number analyzed (Participants) | 136 | 59 | 51
  hSBA-MenA, ≥ 1:8 | 136 | 58 | 8
  hSBA-MenC, ≥ 1:8 | 147 | 66 | 3
  hSBA-MenW-135, ≥ 1:8: number analyzed (Participants) | 107 | 47 | 42
  hSBA-MenW-135, ≥ 1:8 | 107 | 41 | 0
  hSBA-MenY, ≥ 1:8: number analyzed (Participants) | 127 | 52 | 42
  hSBA-MenY, ≥ 1:8 | 127 | 48 | 1

9. Secondary Outcome: hSBA-MenA, hSBA-MenC, hSBA-MenW-135, and hSBA-Men-Y Antibody Titers (One Month Post-primary for Nimenrix 3+1 and Nimenrix 1+1 Groups)) -Randomized Subset of 50% of Subjects of All Three Groups
Description: Antibody titers are presented as geometric mean titers (GMTs).
Time Frame: At Month 5 (one month post-primary for Nimenrix 3+1 and Nimenrix 1+1 Groups)
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Nimenrix 3+1 Group | Nimenrix 1+1 Group | Nimenrix Control Group
Number analyzed (Participants) | 147 | 66 | 59
Titers
  hSBA-MenA: number analyzed (Participants) | 136 | 59 | 51
  hSBA-MenA | 808.0 [683.8 to 954.6] | 270.5 [205.9 to 355.4] | 2.6 [2.2 to 3.1]
  hSBA-MenC | 3970.8 [3144.0 to 5015.1] | 523.1 [381.5 to 717.3] | 2.3 [1.9 to 2.9]
  hSBA-MenW-135: number analyzed (Participants) | 107 | 47 | 42
  hSBA-MenW-135 | 1514.5 [1277.2 to 1795.8] | 136.5 [78.4 to 237.6] | 2.0 [2.0 to 2.0]
  hSBA-MenY: number analyzed (Participants) | 127 | 52 | 42
  hSBA-MenY | 1276.2 [1077.3 to 1511.8] | 194.8 [117.6 to 322.9] | 2.1 [1.9 to 2.4]

10. Secondary Outcome: Number of Participants With hSBA-MenA, hSBA-MenC, hSBA-MenW-135 and hSBA-Men-Y Titers (≥) the Cut-off Value (Pre- and Post-booster for Nimenrix 3+1 and 1+1 Groups and Pre- and Post-vaccination for Nimenrix Control)
Description: The cut-off value for the hSBA titers was ≥ 1:4 and ≥ 1:8.
Time Frame: At Month 13 (pre-booster for Nimenrix 3+1 and Nimenrix 1+1 Groups and pre-vaccination for Nimenrix Control), and at Month 14 (post-booster for Nimenrix 3+1 and Nimenrix 1+1 Groups and post-vaccination for Nimenrix Control)
Population: The analysis was performed on the According-to-Protocol (ATP) cohort for immunogenicity adapted for each timepoint, which included all eligible subjects for whom data concerning immunogenicity endpoint measures were available. The analysis was performed in a randomized subset of 75% of subjects from each group.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix 3+1 Group | Nimenrix 1+1 Group | Nimenrix Control Group
Number analyzed (Participants) | 198 | 92 | 84
Participants
  hSBA-MenA, ≥ 1:4, M13: number analyzed (Participants) | 152 | 71 | 70
  hSBA-MenA, ≥ 1:4, M13 | 131 | 48 | 18
  hSBA-MenA, ≥ 1:4, M14: number analyzed (Participants) | 173 | 83 | 73
  hSBA-MenA, ≥ 1:4, M14 | 173 | 83 | 70
  hSBA-MenC, ≥ 1:4, M13: number analyzed (Participants) | 173 | 78 | 74
  hSBA-MenC, ≥ 1:4, M13 | 168 | 76 | 4
  hSBA-MenC, ≥ 1:4, M14 | 198 | 92 | 84
  hSBA-MenW-135, ≥ 1:4, M13: number analyzed (Participants) | 123 | 53 | 52
  hSBA-MenW-135, ≥ 1:4, M13 | 123 | 53 | 1
  hSBA-MenW-135, ≥ 1:4, M14: number analyzed (Participants) | 129 | 59 | 53
  hSBA-MenW-135, ≥ 1:4, M14 | 129 | 59 | 49
  hSBA-MenY, ≥ 1:4, M13: number analyzed (Participants) | 138 | 61 | 49
  hSBA-MenY, ≥ 1:4, M13 | 137 | 60 | 4
  hSBA-MenY, ≥ 1:4, M14: number analyzed (Participants) | 149 | 69 | 58
  hSBA-MenY, ≥ 1:4, M14 | 149 | 69 | 52
  hSBA-MenA, ≥ 1:8, M13: number analyzed (Participants) | 152 | 71 | 70
  hSBA-MenA, ≥ 1:8, M13 | 130 | 47 | 15
  hSBA-MenA, ≥ 1:8, M14: number analyzed (Participants) | 173 | 83 | 73
  hSBA-MenA, ≥ 1:8, M14 | 173 | 83 | 69
  hSBA-MenC, ≥ 1:8, M13: number analyzed (Participants) | 173 | 78 | 74
  hSBA-MenC, ≥ 1:8, M13 | 168 | 75 | 4
  hSBA-MenC, ≥ 1:8, M14 | 198 | 92 | 84
  hSBA-MenW-135, ≥ 1:8, M13: number analyzed (Participants) | 123 | 53 | 52
  hSBA-MenW-135, ≥ 1:8, M13 | 123 | 53 | 1
  hSBA-MenW-135, ≥ 1:8, M14: number analyzed (Participants) | 129 | 59 | 53
  hSBA-MenW-135, ≥ 1:8, M14 | 129 | 59 | 49
  hSBA-MenY, ≥ 1:8, M13: number analyzed (Participants) | 138 | 61 | 49
  hSBA-MenY, ≥ 1:8, M13 | 137 | 60 | 4
  hSBA-MenY, ≥ 1:8, M14: number analyzed (Participants) | 149 | 69 | 58
  hSBA-MenY, ≥ 1:8, M14 | 149 | 69 | 52

11. Secondary Outcome: hSBA-MenA, hSBA-MenC, hSBA-MenW-135, and hSBA-Men-Y Antibody Titers (Pre-booster for Nimenrix 3+1 and 1+1 Groups and Pre-vaccination for Nimenrix Control, and Post-booster for Nimenrix 3+1 and 1+1 Groups and Post-vaccination for Nimenrix Control)
Description: Antibody titers are presented as geometric mean titers (GMTs).
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Nimenrix 3+1 Group | Nimenrix 1+1 Group | Nimenrix Control Group
Number analyzed (Participants) | 198 | 92 | 84
Titers
  hSBA-MenA, M13: number analyzed (Participants) | 152 | 71 | 70
  hSBA-MenA, M13 | 64.6 [48.8 to 85.5] | 20.8 [13.5 to 32.2] | 3.2 [2.6 to 3.8]
  hSBA-MenA, M14: number analyzed (Participants) | 173 | 83 | 73
  hSBA-MenA, M14 | 2318.6 [1991.7 to 2699.1] | 1415.6 [1140.2 to 1757.5] | 196.3 [140.5 to 274.2]
  hSBA-MenC, M13: number analyzed (Participants) | 173 | 78 | 74
  hSBA-MenC, M13 | 209.0 [165.7 to 263.7] | 150.8 [108.5 to 209.5] | 2.3 [2.0 to 2.7]
  hSBA-MenC, M14 | 15919.1 [13965.3 to 18146.2] | 13360.1 [10952.9 to 16296.4] | 363.3 [269.4 to 490.1]
  hSBA-MenW-135, M13: number analyzed (Participants) | 123 | 53 | 52
  hSBA-MenW-135, M13 | 307.9 [262.9 to 360.6] | 428.6 [328.4 to 559.2] | 2.1 [1.9 to 2.3]
  hSBA-MenW-135, M14: number analyzed (Participants) | 129 | 59 | 53
  hSBA-MenW-135, M14 | 8761.8 [7431.3 to 10330.5] | 9015.6 [7045.2 to 11537.1] | 221.7 [140.6 to 349.5]
  hSBA-MenY, M13: number analyzed (Participants) | 138 | 61 | 49
  hSBA-MenY, M13 | 363.2 [309.9 to 425.7] | 389.2 [292.3 to 518.1] | 2.6 [2.0 to 3.5]
  hSBA-MenY, M14: number analyzed (Participants) | 149 | 69 | 58
  hSBA-MenY, M14 | 5989.3 [5281.0 to 6792.6] | 5977.6 [4746.8 to 7527.6] | 281.5 [171.9 to 460.9]

12. Secondary Outcome: Number of Subjects With Booster Responses for hSBA-MenA, hSBA-MenC, hSBA-MenW-135 and hSBA-MenY in Nimenrix 3+1 and Nimenrix 1+1 Groups and With Vaccine Response in Nimenrix Control Group
Description: Vaccine/Booster response was defined as: for seronegative subjects (rSBA titers < 1:4 pre-vaccination at Month 13), antibody titer ≥ 1:32 at post vaccination; for seropositive subjects (rSBA titers >= 1:4 pre-vaccination at Month 13), antibody titer at post vaccination ≥ 4-fold the pre vaccination.
Time Frame: At Month 14 (one month after the booster dose in Nimenrix 3+1 and Nimenrix 1+1 and post-vaccination in Nimenrix Control Group)
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix 3+1 Group | Nimenrix 1+1 Group | Nimenrix Control Group
Number analyzed (Participants) | 163 | 75 | 65
Participants
  hSBA-MenA, Total: number analyzed (Participants) | 137 | 64 | 58
  hSBA-MenA, Total | 130 | 61 | 51
  hSBA-MenC, Total | 163 | 73 | 65
  hSBA-MenW-135, Total: number analyzed (Participants) | 107 | 42 | 38
  hSBA-MenW-135, Total | 106 | 40 | 37
  hSBA-MenY, Total: number analyzed (Participants) | 122 | 49 | 34
  hSBA-MenY, Total | 115 | 45 | 30

13. Secondary Outcome: Number of Subjects With Anti-pneumococcal Antibody Concentrations Greater Than or Equal to (≥) 0.15 Micrograms Per Milliliter (µg/mL).
Description: The anti-pneumococcal serotypes assessed were 1, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F and 23F.
Time Frame: At Months 5 (one month post-dose 3), Month 13 (prior booster dose) and Month 14 (one month after the booster dose)
Population: The analysis was performed on the According-to-Protocol (ATP) cohort for immunogenicity adapted for each timepoint, which included all eligible subjects for whom data concerning immunogenicity endpoint measures were available. The analysis was performed in a randomized subset of 25% of all subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix 3+1 Group | Nimenrix 1+1 Group | Nimenrix Control Group
Number analyzed (Participants) | 82 | 42 | 37
Participants
  anti-1, M5 | 82 | 42 | 37
  anti-1, M13: number analyzed (Participants) | 57 | 32 | 27
  anti-1, M13 | 36 | 19 | 19
  anti-1, M14: number analyzed (Participants) | 61 | 30 | 29
  anti-1, M14 | 61 | 29 | 29
  anti-4, M5 | 82 | 42 | 37
  anti-4, M13: number analyzed (Participants) | 57 | 33 | 27
  anti-4, M13 | 38 | 22 | 20
  anti-4, M14: number analyzed (Participants) | 61 | 30 | 29
  anti-4, M14 | 61 | 30 | 29
  anti-5, M5 | 81 | 42 | 37
  anti-5, M13: number analyzed (Participants) | 57 | 33 | 27
  anti-5, M13 | 32 | 18 | 17
  anti-5, M14: number analyzed (Participants) | 61 | 30 | 29
  anti-5, M14 | 60 | 29 | 27
  anti-6A, M5: number analyzed (Participants) | 69 | 37 | 28
  anti-6A, M5 | 51 | 31 | 22
  anti-6A, M13: number analyzed (Participants) | 56 | 32 | 26
  anti-6A, M13 | 44 | 26 | 16
  anti-6A, M14: number analyzed (Participants) | 51 | 25 | 25
  anti-6A, M14 | 51 | 25 | 24
  anti-6B, M5: number analyzed (Participants) | 81 | 42 | 37
  anti-6B, M5 | 81 | 41 | 37
  anti-6B, M13: number analyzed (Participants) | 57 | 33 | 27
  anti-6B, M13 | 55 | 31 | 22
  anti-6B, M14: number analyzed (Participants) | 61 | 30 | 29
  anti-6B, M14 | 61 | 30 | 28
  anti-7F, M5 | 82 | 42 | 37
  anti-7F, M13: number analyzed (Participants) | 57 | 33 | 27
  anti-7F, M13 | 55 | 32 | 23
  anti-7F, M14: number analyzed (Participants) | 61 | 30 | 29
  anti-7F, M14 | 61 | 29 | 29
  anti-9V, M5 | 82 | 42 | 37
  anti-9V, M13: number analyzed (Participants) | 57 | 33 | 27
  anti-9V, M13 | 47 | 24 | 17
  anti-9V, M14: number analyzed (Participants) | 61 | 30 | 29
  anti-9V, M14 | 61 | 29 | 29
  anti-14, M5: number analyzed (Participants) | 82 | 42 | 36
  anti-14, M5 | 82 | 42 | 36
  anti-14, M13: number analyzed (Participants) | 57 | 33 | 27
  anti-14, M13 | 56 | 33 | 25
  anti-14, M14: number analyzed (Participants) | 61 | 30 | 29
  anti-14, M14 | 61 | 30 | 29
  anti-18C, M5 | 81 | 42 | 37
  anti-18C, M13: number analyzed (Participants) | 57 | 33 | 27
  anti-18C, M13 | 43 | 20 | 19
  anti-18C, M14: number analyzed (Participants) | 61 | 30 | 29
  anti-18C, M14 | 61 | 29 | 29
  anti-19A, M5 | 49 | 26 | 27
  anti-19A, M13: number analyzed (Participants) | 57 | 33 | 27
  anti-19A, M13 | 41 | 23 | 20
  anti-19A, M14: number analyzed (Participants) | 61 | 29 | 29
  anti-19A, M14 | 57 | 27 | 27
  anti-19F, M5: number analyzed (Participants) | 81 | 42 | 37
  anti-19F, M5 | 81 | 42 | 36
  anti-19F, M13: number analyzed (Participants) | 57 | 33 | 27
  anti-19F, M13 | 57 | 33 | 25
  anti-19F, M14: number analyzed (Participants) | 61 | 30 | 29
  anti-19F, M14 | 61 | 30 | 29
  anti-23F, M5: number analyzed (Participants) | 71 | 42 | 36
  anti-23F, M5 | 66 | 42 | 35
  anti-23F, M13: number analyzed (Participants) | 57 | 33 | 26
  anti-23F, M13 | 42 | 25 | 18
  anti-23F, M14: number analyzed (Participants) | 45 | 24 | 21
  anti-23F, M14 | 45 | 23 | 21

14. Secondary Outcome: Number of Subjects With Anti-pneumococcal Antibody Concentrations Greater Than or Equal to (≥) 0.35 Micrograms Per Milliliter (µg/mL)
Description: The anti-pneumococcal serotypes assessed were 1, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F and 23F.
Time Frame: At Months 5 (one month post-dose 3), Month 13 (prior booster dose) and Month 14 (one month after the booster dose)
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix 3+1 Group | Nimenrix 1+1 Group | Nimenrix Control Group
Number analyzed (Participants) | 82 | 42 | 37
Participants
  anti-1, M5 | 76 | 41 | 34
  anti-1, M13: number analyzed (Participants) | 57 | 32 | 27
  anti-1, M13 | 12 | 5 | 8
  anti-1, M14: number analyzed (Participants) | 61 | 30 | 29
  anti-1, M14 | 61 | 29 | 28
  anti-4, M5 | 81 | 41 | 37
  anti-4, M13: number analyzed (Participants) | 57 | 33 | 27
  anti-4, M13 | 17 | 5 | 10
  anti-4, M14: number analyzed (Participants) | 61 | 30 | 29
  anti-4, M14 | 58 | 29 | 29
  anti-5, M5 | 72 | 32 | 28
  anti-5, M13: number analyzed (Participants) | 57 | 33 | 27
  anti-5, M13 | 10 | 5 | 5
  anti-5, M14: number analyzed (Participants) | 61 | 30 | 29
  anti-5, M14 | 49 | 23 | 26
  anti-6A, M5: number analyzed (Participants) | 69 | 37 | 28
  anti-6A, M5 | 36 | 20 | 13
  anti-6A, M13: number analyzed (Participants) | 56 | 32 | 26
  anti-6A, M13 | 26 | 10 | 11
  anti-6A, M14: number analyzed (Participants) | 51 | 25 | 25
  anti-6A, M14 | 47 | 22 | 23
  anti-6B, M5: number analyzed (Participants) | 81 | 42 | 37
  anti-6B, M5 | 73 | 40 | 35
  anti-6B, M13: number analyzed (Participants) | 57 | 33 | 27
  anti-6B, M13 | 37 | 23 | 15
  anti-6B, M14: number analyzed (Participants) | 61 | 30 | 29
  anti-6B, M14 | 61 | 28 | 28
  anti-7F, M5 | 81 | 42 | 37
  anti-7F, M13: number analyzed (Participants) | 57 | 33 | 27
  anti-7F, M13 | 38 | 17 | 14
  anti-7F, M14: number analyzed (Participants) | 61 | 30 | 29
  anti-7F, M14 | 61 | 29 | 28
  anti-9V, M5 | 79 | 40 | 36
  anti-9V, M13: number analyzed (Participants) | 57 | 33 | 27
  anti-9V, M13 | 19 | 10 | 9
  anti-9V, M14: number analyzed (Participants) | 61 | 30 | 29
  anti-9V, M14 | 59 | 28 | 28
  anti-14, M5: number analyzed (Participants) | 82 | 42 | 36
  anti-14, M5 | 80 | 41 | 36
  anti-14, M13: number analyzed (Participants) | 57 | 33 | 27
  anti-14, M13 | 44 | 28 | 21
  anti-14, M14: number analyzed (Participants) | 61 | 30 | 29
  anti-14, M14 | 61 | 29 | 28
  anti-18C, M5 | 79 | 41 | 36
  anti-18C, M13: number analyzed (Participants) | 57 | 33 | 27
  anti-18C, M13 | 18 | 9 | 11
  anti-18C, M14: number analyzed (Participants) | 61 | 30 | 29
  anti-18C, M14 | 61 | 27 | 29
  anti-19A, M5 | 28 | 14 | 13
  anti-19A, M13: number analyzed (Participants) | 57 | 33 | 27
  anti-19A, M13 | 25 | 15 | 5
  anti-19A, M14: number analyzed (Participants) | 61 | 29 | 29
  anti-19A, M14 | 52 | 21 | 22
  anti-19F, M5: number analyzed (Participants) | 81 | 42 | 37
  anti-19F, M5 | 80 | 42 | 36
  anti-19F, M13: number analyzed (Participants) | 57 | 33 | 27
  anti-19F, M13 | 52 | 30 | 20
  anti-19F, M14: number analyzed (Participants) | 61 | 30 | 29
  anti-19F, M14 | 61 | 30 | 29
  anti-23F, M5: number analyzed (Participants) | 71 | 42 | 36
  anti-23F, M5 | 62 | 42 | 32
  anti-23F, M13: number analyzed (Participants) | 57 | 33 | 26
  anti-23F, M13 | 28 | 14 | 12
  anti-23F, M14: number analyzed (Participants) | 45 | 24 | 21
  anti-23F, M14 | 45 | 23 | 20

15. Secondary Outcome: Anti-pneumococcal Antibody Concentrations
Description: Antibody concentrations were expressed as Geometric Mean Concentrations (GMCs) and measured in micrograms/milliliter (µg/mL)
Time Frame: At Months 5 (one month post-dose 3), Month 13 (prior booster-dose) and Month 14 (one month after the booster dose)
Population: as for outcome 13
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Nimenrix 3+1 Group | Nimenrix 1+1 Group | Nimenrix Control Group
Number analyzed (Participants) | 82 | 42 | 37
μg/mL
  anti-1, M5 | 1.3 [1.1 to 1.6] | 1.4 [1.1 to 1.8] | 1.5 [1.1 to 2.1]
  anti-1, M13: number analyzed (Participants) | 57 | 32 | 27
  anti-1, M13 | 0.2 [0.1 to 0.2] | 0.2 [0.1 to 0.2] | 0.2 [0.2 to 0.3]
  anti-1, M14: number analyzed (Participants) | 61 | 30 | 29
  anti-1, M14 | 2.1 [1.6 to 2.6] | 1.7 [1.2 to 2.5] | 2.2 [1.5 to 3.2]
  anti-4, M5 | 1.7 [1.5 to 2.0] | 1.8 [1.4 to 2.2] | 1.8 [1.3 to 2.5]
  anti-4, M13: number analyzed (Participants) | 57 | 33 | 27
  anti-4, M13 | 0.2 [0.2 to 0.3] | 0.2 [0.2 to 0.3] | 0.3 [0.2 to 0.4]
  anti-4, M14: number analyzed (Participants) | 61 | 30 | 29
  anti-4, M14 | 2.4 [1.8 to 3.1] | 2.4 [1.8 to 3.1] | 3.1 [2.3 to 4.2]
  anti-5, M5 | 0.6 [0.6 to 0.7] | 0.6 [0.5 to 0.7] | 0.7 [0.5 to 0.9]
  anti-5, M13: number analyzed (Participants) | 57 | 33 | 27
  anti-5, M13 | 0.2 [0.1 to 0.2] | 0.2 [0.1 to 0.2] | 0.2 [0.1 to 0.2]
  anti-5, M14: number analyzed (Participants) | 61 | 30 | 29
  anti-5, M14 | 0.7 [0.6 to 0.9] | 0.5 [0.4 to 0.7] | 0.7 [0.5 to 1.0]
  anti-6A, M5: number analyzed (Participants) | 69 | 37 | 28
  anti-6A, M5 | 0.3 [0.3 to 0.4] | 0.4 [0.3 to 0.6] | 0.3 [0.2 to 0.4]
  anti-6A, M13: number analyzed (Participants) | 56 | 32 | 26
  anti-6A, M13 | 0.3 [0.2 to 0.4] | 0.3 [0.2 to 0.4] | 0.2 [0.2 to 0.4]
  anti-6A, M14: number analyzed (Participants) | 51 | 25 | 25
  anti-6A, M14 | 1.7 [1.3 to 2.3] | 1.4 [0.9 to 2.1] | 1.6 [1.0 to 2.5]
  anti-6B, M5: number analyzed (Participants) | 81 | 42 | 37
  anti-6B, M5 | 1.8 [1.4 to 2.3] | 1.7 [1.3 to 2.4] | 1.8 [1.3 to 2.5]
  anti-6B, M13: number analyzed (Participants) | 57 | 33 | 27
  anti-6B, M13 | 0.6 [0.4 to 0.7] | 0.5 [0.4 to 0.7] | 0.4 [0.3 to 0.7]
  anti-6B, M14: number analyzed (Participants) | 61 | 30 | 29
  anti-6B, M14 | 3.8 [3.1 to 4.8] | 2.4 [1.7 to 3.5] | 3.4 [2.2 to 5.2]
  anti-7F, M5 | 2.5 [2.2 to 3.0] | 2.2 [1.8 to 2.7] | 2.8 [2.1 to 3.7]
  anti-7F, M13: number analyzed (Participants) | 57 | 33 | 27
  anti-7F, M13 | 0.4 [0.4 to 0.5] | 0.4 [0.3 to 0.5] | 0.4 [0.3 to 0.6]
  anti-7F, M14: number analyzed (Participants) | 61 | 30 | 29
  anti-7F, M14 | 3.5 [2.9 to 4.2] | 2.2 [1.6 to 3.1] | 3.4 [2.4 to 4.9]
  anti-9V, M5 | 1.2 [1.0 to 1.4] | 1.2 [1.0 to 1.5] | 1.3 [1.0 to 1.7]
  anti-9V, M13: number analyzed (Participants) | 57 | 33 | 27
  anti-9V, M13 | 0.3 [0.2 to 0.4] | 0.3 [0.2 to 0.4] | 0.2 [0.1 to 0.3]
  anti-9V, M14: number analyzed (Participants) | 61 | 30 | 29
  anti-9V, M14 | 1.6 [1.3 to 2.0] | 1.0 [0.8 to 1.4] | 1.6 [1.2 to 2.2]
  anti-14, M5: number analyzed (Participants) | 82 | 42 | 36
  anti-14, M5 | 5.2 [4.1 to 6.5] | 6.0 [4.4 to 8.0] | 7.0 [4.9 to 10.0]
  anti-14, M13: number analyzed (Participants) | 57 | 33 | 27
  anti-14, M13 | 1.0 [0.7 to 1.3] | 0.8 [0.6 to 1.0] | 0.9 [0.5 to 1.4]
  anti-14, M14: number analyzed (Participants) | 61 | 30 | 29
  anti-14, M14 | 8.4 [6.8 to 10.4] | 6.8 [4.8 to 9.7] | 9.0 [6.0 to 13.5]
  anti-18C, M5 | 2.3 [1.9 to 2.8] | 2.0 [1.5 to 2.5] | 2.9 [2.2 to 3.8]
  anti-18C, M13: number analyzed (Participants) | 57 | 33 | 27
  anti-18C, M13 | 0.2 [0.2 to 0.3] | 0.2 [0.1 to 0.3] | 0.3 [0.2 to 0.4]
  anti-18C, M14: number analyzed (Participants) | 61 | 30 | 29
  anti-18C, M14 | 3.6 [3.0 to 4.4] | 2.3 [1.5 to 3.6] | 3.4 [2.6 to 4.6]
  anti-19A, M5 | 0.2 [0.2 to 0.3] | 0.2 [0.2 to 0.4] | 0.2 [0.2 to 0.3]
  anti-19A, M13: number analyzed (Participants) | 57 | 33 | 27
  anti-19A, M13 | 0.3 [0.2 to 0.4] | 0.3 [0.2 to 0.4] | 0.2 [0.1 to 0.3]
  anti-19A, M14: number analyzed (Participants) | 61 | 29 | 29
  anti-19A, M14 | 1.2 [0.8 to 1.7] | 1.1 [0.6 to 1.9] | 0.8 [0.5 to 1.2]
  anti-19F, M5: number analyzed (Participants) | 81 | 42 | 37
  anti-19F, M5 | 3.7 [3.0 to 4.6] | 3.8 [2.7 to 5.3] | 4.7 [3.3 to 6.6]
  anti-19F, M13: number analyzed (Participants) | 57 | 33 | 27
  anti-19F, M13 | 0.9 [0.7 to 1.2] | 0.9 [0.7 to 1.3] | 0.9 [0.5 to 1.5]
  anti-19F, M14: number analyzed (Participants) | 61 | 30 | 29
  anti-19F, M14 | 8.0 [6.2 to 10.2] | 6.9 [4.5 to 10.6] | 9.8 [6.8 to 14.2]
  anti-23F, M5: number analyzed (Participants) | 71 | 42 | 36
  anti-23F, M5 | 1.4 [1.0 to 1.9] | 1.8 [1.4 to 2.4] | 1.5 [1.0 to 2.2]
  anti-23F, M13: number analyzed (Participants) | 57 | 33 | 26
  anti-23F, M13 | 0.3 [0.2 to 0.4] | 0.3 [0.2 to 0.4] | 0.2 [0.2 to 0.4]
  anti-23F, M14: number analyzed (Participants) | 45 | 24 | 21
  anti-23F, M14 | 3.4 [2.6 to 4.5] | 2.1 [1.3 to 3.4] | 2.9 [1.8 to 4.7]

16. Secondary Outcome: Number of Subjects With Anti-diphtheria (Anti-D) Antibodies
Description: Cut-off values assessed were greater than or equal to (≥) 0.1 international units per milliliter (IU/mL).
Time Frame: At Month 5 (one month post-dose 3)
Population: The analysis was performed on a randomized subset of 25% in the primary ATP cohort for immunogenicity who complied with the protocol criteria and for whom data concerning immunogenicity endpoint measures were available, for antibodies against at least one study vaccine antigen component after at least one vaccination during the primary vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix 3+1 Group | Nimenrix 1+1 Group | Nimenrix Control Group
Number analyzed (Participants) | 72 | 34 | 38
Participants | 72 | 34 | 38

17. Secondary Outcome: Concentration of Antibodies Against Diphtheria Antigens (Anti-D)
Description: Concentrations are presented as geometric mean concentrations (GMCs) expressed in international units per milliliter (IU/mL).
Time Frame: At Month 5 (one month post-dose 3)
Population: as for outcome 16
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Nimenrix 3+1 Group | Nimenrix 1+1 Group | Nimenrix Control Group
Number analyzed (Participants) | 72 | 34 | 38
IU/mL | 2.259 [1.820 to 2.804] | 3.028 [2.177 to 4.213] | 2.462 [1.700 to 3.565]

18. Secondary Outcome: Concentration of Antibodies Against Diphtheria Antigens (Anti-D)
Description: Concentrations are presented as geometric mean concentrations (GMCs) expressed in international units per milliliter (IU/mL). The analysis was performed in a randomized subset of 25% of subjects of all three groups. Note: As the percentage of subjects with serological results excluded from the ATP cohorts was higher than 5%, a second analysis based on the total vaccinated cohorts (TVCs) (Primary and Booster) was performed to complement the ATP analysis.
Time Frame: At Month 5 (one month post-dose 3)
Population: The analysis was performed on the Primary TVC, which included all vaccinated subjects during the primary phase.
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Nimenrix 3+1 Group | Nimenrix 1+1 Group | Nimenrix Control Group
Number analyzed (Participants) | 76 | 36 | 39
IU/mL | 2.435 [1.958 to 3.028] | 3.069 [2.225 to 4.233] | 2.423 [1.688 to 3.479]

19. Secondary Outcome: Concentration of Antibodies Against Pertussis Toxoid (Anti-PT), Filamentous Haemagglutinin (Anti-FHA), Pertactin (Anti-PRN) Antigens
Description: Concentrations are presented as geometric mean concentrations (GMCs) expressed in enzyme-linked immunosorbent assay (ELISA) units per milliliter (EL.U/ml).
Time Frame: At Month 5 (one month post-dose 3)
Population: as for outcome 16
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Nimenrix 3+1 Group | Nimenrix 1+1 Group | Nimenrix Control Group
Number analyzed (Participants) | 73 | 34 | 39
EL.U/mL
  anti-PT, M5 | 49.9 [43.3 to 57.6] | 51.9 [40.8 to 66.0] | 47.8 [38.3 to 59.7]
  anti-FHA, M5 | 126.2 [108.8 to 146.3] | 134.2 [108.3 to 166.4] | 132.6 [107.8 to 163.1]
  anti-PRN, M5 | 108.6 [88.8 to 132.9] | 167.5 [117.6 to 238.7] | 158.2 [106.5 to 235.1]

20. Secondary Outcome: Number of Subjects With Anti-pertussis Toxoid (Anti-PT), Anti-filamentous Haemagglutinin (Anti-FHA), Anti-pertactin (Anti-PRN) Immunoglobulin G (IgG) Antibodies
Description: Cut-off values assessed were greater than or equal to ≥ 5 enzyme-linked immunosorbent assay (ELISA) units per milliliter (EL.U/ml).
Time Frame: At Month 5 (one month post-dose 3)
Population: The analysis was performed on the Primary TVC included all vaccinated subjects during the primary phase.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix 3+1 Group | Nimenrix 1+1 Group | Nimenrix Control Group
Number analyzed (Participants) | 77 | 36 | 40
Participants
  anti-PT, M5 | 77 | 36 | 40
  anti-FHA, M5 | 77 | 36 | 40
  anti-PRN, M5 | 77 | 36 | 39

21. Secondary Outcome: Concentration of Antibodies Against Pertussis Toxoid (Anti-PT), Filamentous Haemagglutinin (Anti-FHA), Pertactin (Anti-PRN) Antigens
Description: as for outcome 19
Time Frame: At Month 5 (one month post-dose 3)
Population: The analysis was performed on the Primary TVC, which included all vaccinated subjects during the primary phase.
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Nimenrix 3+1 Group | Nimenrix 1+1 Group | Nimenrix Control Group
Number analyzed (Participants) | 77 | 36 | 40
EL.U/mL
  anti-PT, M5 | 50.4 [43.9 to 57.8] | 54.7 [42.9 to 69.9] | 46.4 [37.0 to 58.1]
  anti-FHA, M5 | 127.3 [110.6 to 146.6] | 143.3 [114.4 to 179.4] | 129.4 [105.1 to 159.2]
  anti-PRN, M5 | 116.7 [95.2 to 143.1] | 178.9 [125.5 to 255.1] | 154.8 [105.0 to 228.3]

22. Secondary Outcome: Antibody Titers for Anti-polio Type 1, 2 and 3 Antibodies
Description: Antibody titers are presented as geometric mean titers (GMTs).
Time Frame: At Month 5 (one month post-dose 3)
Population: as for outcome 16
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Nimenrix 3+1 Group | Nimenrix 1+1 Group | Nimenrix Control Group
Number analyzed (Participants) | 69 | 29 | 33
Titers
  anti-Polio 1, M5: number analyzed (Participants) | 69 | 28 | 29
  anti-Polio 1, M5 | 788.8 [584.1 to 1065.2] | 1102.9 [725.2 to 1677.2] | 908.6 [549.1 to 1503.4]
  anti-Polio 2, M5 | 850.4 [647.3 to 1117.3] | 953.3 [579.0 to 1569.5] | 1079.2 [704.9 to 1652.1]
  anti-Polio 3, M5: number analyzed (Participants) | 68 | 26 | 30
  anti-Polio 3, M5 | 1678.8 [1211.2 to 2326.9] | 1676.7 [1011.1 to 2780.5] | 1261.3 [720.8 to 2207.1]

23. Secondary Outcome: Antibody Titers for Anti-polio Type 1, 2 and 3 Antibodies
Description: Antibody titers are presented as geometric mean titers (GMTs). The analysis was performed in a randomized subset of 25% of subjects of all three groups. Note: As the percentage of subjects with serological results excluded from the ATP cohorts was higher than 5%, a second analysis based on the total vaccinated cohorts (TVCs) (Primary and Booster) was performed to complement the ATP analysis.
Time Frame: At Month 5 (one month post-dose 3)
Population: The analysis was performed on the Primary TVC, which included all vaccinated subjects during the primary phase.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Nimenrix 3+1 Group | Nimenrix 1+1 Group | Nimenrix Control Group
Number analyzed (Participants) | 73 | 31 | 34
Titers
  anti-Polio 1, M5: number analyzed (Participants) | 73 | 30 | 30
  anti-Polio 1, M5 | 827.2 [618.7 to 1105.8] | 1048.1 [681.1 to 1612.7] | 861.0 [523.3 to 1416.8]
  anti-Polio 2, M5 | 931.3 [707.7 to 1225.6] | 990.4 [606.5 to 1617.3] | 1024.0 [668.6 to 1568.2]
  anti-Polio 3, M5: number analyzed (Participants) | 71 | 28 | 31
  anti-Polio 3, M5 | 1709.5 [1245.4 to 2346.7] | 1618.7 [963.7 to 2719.0] | 1184.8 [679.9 to 2064.4]

24. Secondary Outcome: Number of Subjects With Anti-tetanus (Anti-T) Antibodies
Description: Cut-off values assessed were greater than or equal to (≥) 0.1 international units per milliliter (IU/mL).
Time Frame: At Months 5 (one month post-dose 3), Month 13 (prior booster-dose) and Month 14 (one month after the booster dose)
Population: The analysis was performed on the ATP cohort for immunogenicity adapted for each timepoint, which included all eligible subjects, who complied with the vaccination schedule and for whom data concerning immunogenicity endpoint measures were available. The analysis was performed in a randomized subset of 25% of subjects of all three groups.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix 3+1 Group | Nimenrix 1+1 Group | Nimenrix Control Group
Number analyzed (Participants) | 77 | 36 | 40
Participants
  anti-T, M5 | 77 | 36 | 40
  anti-T, M13: number analyzed (Participants) | 59 | 29 | 26
  anti-T, M13 | 58 | 28 | 24
  anti-T, M14: number analyzed (Participants) | 62 | 22 | 23
  anti-T, M14 | 62 | 22 | 23

25. Secondary Outcome: Concentration of Antibodies Against Tetanus Antigens (Anti-T)
Description: as for outcome 17
Time Frame: At Months 5 (one month post-dose 3), Month 13 (prior booster-dose) and Month 14 (one month after the booster dose)
Population: as for outcome 24
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Nimenrix 3+1 Group | Nimenrix 1+1 Group | Nimenrix Control Group
Number analyzed (Participants) | 73 | 34 | 39
IU/mL
  anti-T, M5 | 5.798 [4.998 to 6.726] | 7.246 [5.305 to 9.897] | 5.973 [4.818 to 7.406]
  anti-T, M13: number analyzed (Participants) | 49 | 24 | 21
  anti-T, M13 | 0.479 [0.398 to 0.576] | 0.659 [0.427 to 1.018] | 0.461 [0.297 to 0.716]
  anti-T, M14: number analyzed (Participants) | 57 | 20 | 21
  anti-T, M14 | 18.977 [16.013 to 22.489] | 16.813 [12.386 to 22.821] | 35.835 [23.802 to 53.951]

26. Secondary Outcome: Number of Subjects With Anti-tetanus (Anti-T) Antibodies
Description: Cut-off values assessed were greater than or equal to (≥) 0.1 international units per milliliter (IU/mL). The analysis was performed in a randomized subset of 25% of subjects of all three groups. Note: As the percentage of subjects with serological results excluded from the ATP cohorts was higher than 5%, a second analysis based on the total vaccinated cohorts (TVCs) (Primary and Booster) was performed to complement the ATP analysis.
Time Frame: At Months 5 (one month post-dose 3), 13 (prior booster-dose) and 14 (one month after the booster dose)
Population: The analysis was performed on the Adapted TVC, which included all vaccinated subjects during the primary phase.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix 3+1 Group | Nimenrix 1+1 Group | Nimenrix Control Group
Number analyzed (Participants) | 77 | 36 | 40
Participants
  anti-T, M5 | 77 | 36 | 40
  anti-T, M13: number analyzed (Participants) | 59 | 29 | 26
  anti-T, M13 | 58 | 28 | 24
  anti-T, 14: number analyzed (Participants) | 62 | 22 | 23
  anti-T, 14 | 62 | 22 | 23

27. Secondary Outcome: Anti-PRP Antibody Concentrations (Geometric Mean Concentrations) in a Randomized Subset of 25% of the Subjects
Description: The endpoints evaluating immunogenicity of the Hib component (anti-polyribosyl ribitol phosphate [anti-PRP] antibody concentrations) has been cancelled owing to the extended delay in the re-development and re-validation of the PRP assay.
Time Frame: At Month 5 (one month post-dose 3)
Population: No subjects were analyzed because the endpoints evaluating immunogenicity of the Hib component (anti-polyribosyl ribitol phosphate [anti-PRP] antibody concentrations) has been cancelled owing to the extended delay in the re-development and re-validation of the PRP assay.
Arm/Group | Nimenrix 3+1 Group | Nimenrix 1+1 Group | Nimenrix Control Group
Number analyzed (Participants) | 0 | 0 | 0

28. Secondary Outcome: Number of Subjects With Solicited Local Symptoms (Primary Phase)
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = pain that prevented normal activity. Grade 3 redness/swelling = redness/swelling spreading beyond 30 millimeters (mm) of injection site.
Time Frame: Within 8 days (Day 0-7) post primary vaccination
Population: The analysis was performed on the Primary Total Vaccinated cohort, which included all vaccinated subjects during the primary phase who had their symptom sheets completed.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix 3+1 Group | Nimenrix 1+1 Group | Nimenrix Control Group
Number analyzed (Participants) | 369 | 182 | 184
Participants
  Any Pain Dose 1 | 220 | 115 | 108
  Grade 3 Pain Dose 1 | 38 | 25 | 14
  Any Redness Dose 1 | 94 | 39 | 43
  Grade 3 Redness Dose 1 | 1 | 0 | 0
  Any Swelling Dose 1 | 84 | 31 | 34
  Grade 3 Swelling Dose 1 | 0 | 3 | 0
  Any Pain Dose 2: number analyzed (Participants) | 363 | 181 | 181
  Any Pain Dose 2 | 177 | 92 | 101
  Grade 3 Pain Dose 2: number analyzed (Participants) | 363 | 181 | 181
  Grade 3 Pain Dose 2 | 33 | 11 | 16
  Any Redness Dose 2: number analyzed (Participants) | 363 | 181 | 181
  Any Redness Dose 2 | 93 | 51 | 48
  Grade 3 Redness Dose 2: number analyzed (Participants) | 363 | 181 | 181
  Grade 3 Redness Dose 2 | 2 | 0 | 1
  Any Swelling Dose 2: number analyzed (Participants) | 363 | 181 | 181
  Any Swelling Dose 2 | 76 | 47 | 42
  Grade 3 Swelling Dose 2: number analyzed (Participants) | 363 | 181 | 181
  Grade 3 Swelling Dose 2 | 2 | 2 | 0
  Any Pain Dose 3: number analyzed (Participants) | 359 | 177 | 180
  Any Pain Dose 3 | 148 | 73 | 93
  Grade 3 Pain Dose 3: number analyzed (Participants) | 359 | 177 | 180
  Grade 3 Pain Dose 3 | 16 | 18 | 9
  Any Redness Dose 3: number analyzed (Participants) | 359 | 177 | 180
  Any Redness Dose 3 | 74 | 46 | 42
  Grade 3 Redness Dose 3: number analyzed (Participants) | 359 | 177 | 180
  Grade 3 Redness Dose 3 | 1 | 1 | 1
  Any Swelling Dose 3: number analyzed (Participants) | 359 | 177 | 180
  Any Swelling Dose 3 | 66 | 46 | 37
  Grade 3 Swelling Dose 3: number analyzed (Participants) | 359 | 177 | 180
  Grade 3 Swelling Dose 3 | 1 | 0 | 0
  Any Pain Across Doses | 262 | 135 | 142
  Grade 3 Pain Across Doses | 65 | 36 | 33
  Any Redness Across Doses | 160 | 79 | 78
  Grade 3 Redness Across Doses | 4 | 1 | 2
  Any Swelling Across Doses | 147 | 74 | 70
  Grade 3 Swelling Across Doses | 3 | 4 | 0

29. Secondary Outcome: Number of Subjects With Solicited Local Symptoms (Booster Phase)
Description: as for outcome 28
Time Frame: Within 8 days (Day 0-7) post booster vaccination
Population: The analysis was performed on the Booster Total Vaccinated cohort, which included all vaccinated subjects at booster time point (at Month 13) who had their symptom sheets completed.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix 3+1 Group | Nimenrix 1+1 Group | Nimenrix Control Group
Number analyzed (Participants) | 338 | 165 | 167
Participants
  Any Pain | 139 | 71 | 77
  Grade 3 Pain | 21 | 19 | 14
  Any Redness | 74 | 32 | 39
  Grade 3 Redness | 1 | 1 | 3
  Any Swelling | 55 | 29 | 33
  Grade 3 Swelling | 2 | 1 | 3

30. Secondary Outcome: Number of Subjects With Solicited General Symptoms (Primary Phase)
Description: Assessed solicited general symptoms were temperature [defined as rectally temperature equal to or above 38 degrees Celsius (°C)], drowsiness, irritability and loss of appetite. Any = occurrence of the symptom regardless of intensity grade. Grade 3 symptom = symptom that prevented normal activity. Grade 3 temperature = temperature > 40.0 °C. Related = symptom assessed by the investigator as related to the vaccination.
Time Frame: Within 8 days (Day 0-7) post primary vaccination
Population: as for outcome 28
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix 3+1 Group | Nimenrix 1+1 Group | Nimenrix Control Group
Number analyzed (Participants) | 369 | 182 | 184
Participants
  Any Drowsiness Dose 1 | 177 | 93 | 84
  Grade 3 Drowsiness Dose 1 | 18 | 10 | 2
  Related Drowsiness Dose 1 | 160 | 84 | 79
  Any Irritability Dose 1 | 200 | 107 | 99
  Grade 3 Irritability Dose 1 | 19 | 9 | 10
  Related Irritability Dose 1 | 188 | 96 | 89
  Any Loss of appetite Dose 1 | 109 | 62 | 42
  Grade 3 Loss of appetite Dose 1 | 7 | 5 | 3
  Related Loss of appetite Dose 1 | 99 | 55 | 35
  Any Temperature Dose 1 | 126 | 62 | 58
  Grade 3 Temperature Dose 1 | 0 | 0 | 1
  Related Temperature Dose 1 | 109 | 56 | 53
  Any Drowsiness Dose 2: number analyzed (Participants) | 363 | 181 | 181
  Any Drowsiness Dose 2 | 116 | 72 | 67
  Grade 3 Drowsiness Dose 2: number analyzed (Participants) | 363 | 181 | 181
  Grade 3 Drowsiness Dose 2 | 9 | 8 | 8
  Related Drowsiness Dose 2: number analyzed (Participants) | 363 | 181 | 181
  Related Drowsiness Dose 2 | 109 | 69 | 62
  Any Irritability Dose 2: number analyzed (Participants) | 363 | 181 | 181
  Any Irritability Dose 2 | 163 | 82 | 90
  Grade 3 Irritability Dose 2: number analyzed (Participants) | 363 | 181 | 181
  Grade 3 Irritability Dose 2 | 20 | 14 | 10
  Related Irritability Dose 2: number analyzed (Participants) | 363 | 181 | 181
  Related Irritability Dose 2 | 158 | 77 | 85
  Any Loss of appetite Dose 2: number analyzed (Participants) | 363 | 181 | 181
  Any Loss of appetite Dose 2 | 89 | 50 | 44
  Grade 3 Loss of appetite Dose 2: number analyzed (Participants) | 363 | 181 | 181
  Grade 3 Loss of appetite Dose 2 | 6 | 5 | 6
  Related Loss of appetite Dose 2: number analyzed (Participants) | 363 | 181 | 181
  Related Loss of appetite Dose 2 | 80 | 48 | 39
  Any Temperature Dose 2: number analyzed (Participants) | 363 | 181 | 181
  Any Temperature Dose 2 | 119 | 64 | 63
  Grade 3 Temperature Dose 2: number analyzed (Participants) | 363 | 181 | 181
  Grade 3 Temperature Dose 2 | 0 | 0 | 0
  Related Temperature Dose 2: number analyzed (Participants) | 363 | 181 | 181
  Related Temperature Dose 2 | 116 | 59 | 54
  Any Drowsiness Dose 3: number analyzed (Participants) | 359 | 177 | 180
  Any Drowsiness Dose 3 | 102 | 54 | 64
  Grade 3 Drowsiness Dose 3: number analyzed (Participants) | 359 | 177 | 180
  Grade 3 Drowsiness Dose 3 | 11 | 8 | 4
  Related Drowsiness Dose 3: number analyzed (Participants) | 359 | 177 | 180
  Related Drowsiness Dose 3 | 95 | 54 | 60
  Any Irritability Dose 3: number analyzed (Participants) | 359 | 177 | 180
  Any Irritability Dose 3 | 140 | 73 | 73
  Grade 3 Irritability Dose 3: number analyzed (Participants) | 359 | 177 | 180
  Grade 3 Irritability Dose 3 | 14 | 14 | 3
  Related Irritability Dose 3: number analyzed (Participants) | 359 | 177 | 180
  Related Irritability Dose 3 | 132 | 72 | 69
  Any Loss of appetite Dose 3: number analyzed (Participants) | 359 | 177 | 180
  Any Loss of appetite Dose 3 | 76 | 43 | 50
  Grade 3 Loss of appetite Dose 3: number analyzed (Participants) | 359 | 177 | 180
  Grade 3 Loss of appetite Dose 3 | 7 | 6 | 3
  Related Loss of appetite Dose 3: number analyzed (Participants) | 359 | 177 | 180
  Related Loss of appetite Dose 3 | 63 | 41 | 46
  Any Temperature Dose 3: number analyzed (Participants) | 359 | 177 | 180
  Any Temperature Dose 3 | 109 | 51 | 41
  Grade 3 Temperature Dose 3: number analyzed (Participants) | 359 | 177 | 180
  Grade 3 Temperature Dose 3 | 2 | 0 | 0
  Related Temperature Dose 3: number analyzed (Participants) | 359 | 177 | 180
  Related Temperature Dose 3 | 96 | 46 | 36
  Any Drowsiness Across Doses | 217 | 121 | 118
  Grade 3 Drowsiness Across Doses | 30 | 19 | 13
  Related Drowsiness Across Doses | 205 | 116 | 114
  Any Irritability Across Doses | 254 | 128 | 126
  Grade 3 Irritability Across Doses | 42 | 27 | 18
  Related Irritability Across Doses | 246 | 125 | 121
  Any Loss of appetite Across | 165 | 89 | 82
  Grade 3 Loss of appetite Across | 17 | 13 | 10
  Related Loss of appetite Across | 151 | 84 | 77
  Any Temperature Across Doses | 203 | 102 | 101
  Grade 3 Temperature Across Doses | 2 | 0 | 1
  Related Temperature Across Doses | 193 | 97 | 93

31. Secondary Outcome: Number of Subjects With Solicited General Symptoms (Booster Phase)
Description: as for outcome 30
Time Frame: Within 8 days (Day 0-7) post booster vaccination
Population: as for outcome 29
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix 3+1 Group | Nimenrix 1+1 Group | Nimenrix Control Group
Number analyzed (Participants) | 338 | 165 | 167
Participants
  Any Drowsiness | 79 | 46 | 43
  Grade 3 Drowsiness | 4 | 7 | 5
  Related Drowsiness | 75 | 42 | 43
  Any Irritability | 112 | 54 | 61
  Grade 3 Irritability | 9 | 12 | 10
  Related Irritability | 106 | 52 | 60
  Any Loss of appetite | 69 | 37 | 39
  Grade 3 Loss of appetite | 5 | 5 | 1
  Related Loss of appetite | 60 | 34 | 37
  Any Temperature | 68 | 35 | 27
  Grade 3 Temperature | 2 | 1 | 0
  Related Temperature | 62 | 32 | 24

32. Secondary Outcome: Number of Subjects With Unsolicited Adverse Events (AEs) (Primary Phase)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination.
Time Frame: Within 31 days (Day 0-30) post each primary vaccine dose
Population: The analysis was performed on the Primary Total Vaccinated cohort, which included all vaccinated subjects during the primary phase.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix 3+1 Group | Nimenrix 1+1 Group | Nimenrix Control Group
Number analyzed (Participants) | 376 | 187 | 187
Participants
  Any AE(s) Dose 1 | 67 | 36 | 34
  Any AE(s) Dose 2: number analyzed (Participants) | 368 | 182 | 182
  Any AE(s) Dose 2 | 70 | 34 | 28
  Any AE(s) Dose 3: number analyzed (Participants) | 362 | 179 | 181
  Any AE(s) Dose 3 | 97 | 49 | 45

33. Secondary Outcome: Number of Subjects With Unsolicited Adverse Events (AEs) (Booster Phase)
Description: as for outcome 32
Time Frame: Within 31 days (Day 0-30) post booster vaccination
Population: The analysis was performed on the Booster Total Vaccinated cohort, which included all vaccinated subjects at booster time point (at Month 13).
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix 3+1 Group | Nimenrix 1+1 Group | Nimenrix Control Group
Number analyzed (Participants) | 342 | 166 | 170
Participants | 58 | 32 | 36

34. Secondary Outcome: Number of Subjects With New Onset of Chronic Illnesses (NOCIs)
Description: NOCIs include autoimmune disorders, asthma, type I diabetes, allergies.
Time Frame: From Day 0 to Month 19
Population: as for outcome 32
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix 3+1 Group | Nimenrix 1+1 Group | Nimenrix Control Group
Number analyzed (Participants) | 376 | 187 | 187
Participants | 16 | 8 | 4

35. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: From Day 0 to Month 19
Population: as for outcome 32
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix 3+1 Group | Nimenrix 1+1 Group | Nimenrix Control Group
Number analyzed (Participants) | 376 | 187 | 187
Participants | 35 | 14 | 14

ADVERSE EVENTS:
Time Frame: Solicited local/general symptoms during the 8-day post-vaccination period (Days 0-7), Unsolicited AEs during the 31-day post-vaccination (Days 0-30), SAEs during the entire study period (Day 0 - Month 19).
Arm/Group | Nimenrix 3+1 Group | Nimenrix 1+1 Group | Nimenrix Control Group
All-Cause Mortality (participants affected / at risk) | 0/376 | 0/187 | 1/187
Serious Adverse Events (participants affected / at risk) | 35/376 | 14/187 | 14/187
Other Adverse Events (participants affected / at risk) | 334/376 | 169/187 | 169/187
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nimenrix 3+1 Group (N=376) | Nimenrix 1+1 Group (N=187) | Nimenrix Control Group (N=187)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1)
Ileus paralytic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Sudden infant death syndrome (General disorders) | 0 (0) | 0 (0) | 1 (1)
Anaphylactic shock (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 1 (2) | 0 (0)
Milk allergy (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Amoebic dysentery (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bronchiolitis (Infections and infestations) | 5 (7) | 1 (1) | 3 (3)
Bronchitis (Infections and infestations) | 3 (3) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Escherichia urinary tract infection (Infections and infestations) | 1 (2) | 2 (2) | 0 (0)
Gastroenteritis (Infections and infestations) | 4 (4) | 1 (1) | 3 (3)
Gastroenteritis rotavirus (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
Measles (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Neurological infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Pharyngotonsillitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 13 (16) | 2 (2) | 3 (3)
Pneumonia viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Roseola (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 2 (2) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Burns first degree (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Burns second degree (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Foreign body (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Skull fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 1 (1)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Febrile convulsion (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Hyponatraemic seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 1 (2)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nimenrix 3+1 Group (N=376) | Nimenrix 1+1 Group (N=187) | Nimenrix Control Group (N=187)
Cough (Respiratory, thoracic and mediastinal disorders) | 23 (25) | 8 (8) | 5 (5)
Decreased appetite (Metabolism and nutrition disorders) | 185 (343) | 95 (192) | 95 (175)
Diarrhoea (Gastrointestinal disorders) | 36 (38) | 15 (16) | 10 (10)
Erythema (Skin and subcutaneous tissue disorders) | 177 (335) | 87 (168) | 87 (172)
Irritability (Psychiatric disorders) | 262 (616) | 130 (316) | 130 (323)
Nasopharyngitis (Infections and infestations) | 65 (83) | 27 (42) | 26 (35)
Pain (General disorders) | 273 (684) | 142 (351) | 145 (379)
Pharyngitis (Infections and infestations) | 39 (42) | 17 (25) | 27 (32)
Pyrexia (General disorders) | 215 (426) | 112 (214) | 111 (192)
Somnolence (Nervous system disorders) | 224 (475) | 124 (265) | 120 (258)
Swelling (General disorders) | 157 (281) | 83 (153) | 78 (146)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.